CLINICAL TRIAL: NCT06459830
Title: Effects of Mime Therapy With and Without Neural Mobilization on Facial Symmetry, Synkinesis and Functional Abilities in Patients With Bell's Palsy.
Brief Title: Mime Therapy With and Without Neural Mobilization in Bell's Palsy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0272
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Bell Palsy
Keywords: Bell's palsy; Facial Asymmetry; Facial Paralysis; Mime therapy; Mobilization
MeSH Terms: conditions — Bell Palsy; Facial Asymmetry; Facial Paralysis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mime Therapy with Neural Mobilization (Experimental): This group will receive mime therapy and neural mobilization session with resting intervals.
  1. Self- facial massages for 10 minutes.
  2. Breathing and relaxation exercises .
  3. Exercises to enhance coordination between both sides of the face and to reduce synkinesis.
  4. Exercises to assist with eye and lip closure.
  5. Articulation Exercises.
  6. Facial expression exercises
  Facial Nerve Mobilization The circular movement and horizontal traction will be applied 25 times in three sets with a 5-second rest period in between a single manipulation and a 30- second rest period in between the sets.
  All the participates in the experimental group will receive 15 treatment sessions. Each session will held for 60 minutes per day, 5 days per week, for total duration of 3 weeks.
  Interventions: Other: Mime Therapy with Neural Mobilization
- Mime Therapy with placebo Mobilization (Placebo Comparator): Control group will receive mime therapy session with short resting intervals.
  1. Self- facial massages for 10 minutes.
  2. Breathing and relaxation exercises.
  3. Exercises to enhance coordination between both sides of the face and to reduce synkinesis.
  4. Exercises to assist with eye and lip closure.
  5. Articulation Exercises.
  6. Facial expression exercises.
  Placebo Neural Mobilization Technique:
  Placebo Mobilization followed all the procedures of real facial mobilization without applying horizontal and circular auricular traction. The purpose of this placebo facial nerve mobilization is not to deprived the control group from therapy.
  All the participates in the control group will receive 15 treatment sessions. Each session will held for 60 minutes per day, 5 days per week, for total duration of 3 weeks.
  Interventions: Other: Mime Therapy with Placebo Mobilization

INTERVENTIONS:
Other: Mime Therapy with Neural Mobilization — Experimental group will receive mime therapy and neural mobilization session with small resting intervals.
  Self- facial massages for 10 minutes. Breathing and relaxation exercises for 5 mins. Exercises to enhance coordination between both sides of the face and to reduce synkinesis.
  Exercises to assist with eye and lip closure for 5 mins. Articulation Exercises for 5 mins. Facial expression exercises for 10 mins.
  Facial Neural Mobilization:
  Facial mobilization technique will apply when the patient in supine position with head on the table in neural rotation.
  The circular movement and horizontal traction will be applied 25 times in three sets with a 5-second rest period in between a single manipulation and a 30- second rest period in between the sets.
  All the participates in the experimental group will receive 15 treatment sessions. Each session will held for 60 minutes per day, 5 days per week, for total duration of 3 weeks.
  Arms: Mime Therapy with Neural Mobilization
Other: Mime Therapy with Placebo Mobilization — Control group will receive mime therapy and placebo nerve mobilization session with small resting intervals.
  Self- facial massages for 10 minutes. Breathing and relaxation exercises for 5 mins. Exercises to enhance coordination between both sides of the face and to reduce synkinesis.
  Exercises to assist with eye and lip closure for 5 mins. Articulation Exercises for 5 mins. Facial expression exercises for 10 mins.
  Placebo Nerve Mobilization Technique:
  The placebo nerve mobilization followed all the procedures of real nerve mobilization without applying horizontal and circular auricular traction. The purpose of this placebo nerve mobilization is not to deprived the control group from therapy and equalize the time duration of treatment protocol.
  All the participates in the control group will receive 15 treatment sessions. Each session will held for 60 minutes per day, 5 days per week, for total duration of 3 weeks.
  Arms: Mime Therapy with placebo Mobilization

SUMMARY:
To determine the Effects of Mime Therapy with and without Neural Mobilization on Facial symmetry, Synkinesis and Functional abilities in Patients with Bell's Palsy.

It has been proven that Mime therapy is effective on activating muscles through articulation exercises, facial expression exercises, breathing exercises and facial massages which can alleviate synkinesis, enhance facial symmetry and promote facial functional abilities. On the other hand, facial neural mobilization has recently reported as a safe and effective adjunctive therapy for patients with Bell's palsy due to the facilitation of nerve gliding in the canal impacts by reducing nerve adherence dispersion of noxious inflammatory agents and increasing neural blood supply. So, by incorporating the Neural mobilization with Mime therapy, therapist may enhance overall facial symmetry, reduce the strain on the facial muscles and alleviate synkinesis. So, it may prove to be an upgraded treatment option for clinicians.

DETAILED DESCRIPTION:
A randomized controlled trail conducted in 2023, to evaluate the effect of facial neural mobilization over conventional therapy in improving facial symmetry in patients with acute Bell's palsy. The intervention included 10 days of drug therapy including 3 weeks of conventional therapy to the experimental and the control group. However, the experimental group received additional nerve mobilization technique aimed at mobilizing the facial nerve at the origin of external auditory meatus. Facial neural mobilization is likely to be an effective adjunctive intervention in addition to conventional therapy in improving facial symmetry in acute Bell's palsy.

Randomized clinical trial in 2021 aims to compare the effectiveness of mime therapy and neuromuscular re-education in improving facial symmetry and function in patients with acute Bell's palsy. Both mime therapy and neuromuscular re-education showed highly significant improvements within each group for both outcomes; they showed no difference between each group for the Sunnybrook Facial Grading System (P=0.212) and Facial Clinimetric Evaluation Scale (P=0.97). Both techniques are equally effective in the recovery of facial symmetry and function in acute Bell's palsy.

Another Author conducted a comparative interventional study in 2020 to compare the effects of Electromyography Biofeedback (EMG BFB) and Mime Therapy on electrophysiological parameters in subjects with Bell's palsy. A group of 31 subjects were selected for the study. Conventional physiotherapy with an EMG BFB and Mime therapy has an equal positive effect on electrophysiological parameters in subjects with Bell's palsy.

Many existing studies highlight the impact of Mime therapy on bell's palsy and related outcomes such as facial symmetry, synkinesis and functional abilities. Also, neural mobilization is reported as a safe and effective adjunctive therapy for patients with Bell's palsy. However, up to the researcher's knowledge, there is no research specifically on combined effects of Mime therapy and neural mobilization in patients with bell's palsy. So, this study aims to bridge this gap by investigating these effects. Moreover, it may help the clinicians to have an upgraded approach to treat these patients.

ELIGIBILITY:
Inclusion Criteria:

Idiopathic bell's palsy. Age between 20 to 40 years. Both genders Sub-acute Bell's palsy lasting 3-6 months. Unilateral loss of facial weakness Intact taste sensation. House Brackman grade 4 and 5 (moderate to severe Bell's palsy)

Exclusion Criteria:

Facial palsy recurrence. Patients with Diabetes, Hypertension, and any Auto-immune disorder. Chronic bell's palsy patients Patients with upper motor neuron lesions. Other cranial nerves problem. Pregnancy. Dental metal prosthesis. Facial surgery Skin allergy on face. Patients with Ear infection. Patients with Ear implants. Any neuro-degenerative disorder. Patients with Herpes zoster, Otitis media and Ramsay Hunt syndrome

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Sunny brook facial grading system | 3rd week
  Facial symmetry was measured using the 13-item SFGS. The system includes three components: resting symmetry, the symmetry of voluntary movements, and synkinesis.
  A composite facial symmetry score is calculated as [4 × symmetry of voluntary movement - 5 × resting asymmetry + 1 × synkinesis] with 100 representing normal facial symmetry.
  The SFGS is as reliable when applied by novice users as by expert users. Researchers are using this method more frequently because it has been demonstrated to be repeatable, to have minimal inter-observer and intra-observer variability, and to be responsive to changes over time and as a consequence to treatments. The SFGS has high reliability and repeatability which is good to excellent ranging from 0.766 to 0.860.
Facial disability index | 3rd week
  The FDI helps to measure the difficulties of the face in activities of daily living such as eating, drinking, and communicating. It represents the relationship between impairments, disability, and psychosocial status and also focuses on the disability of individuals with disorders of the facial motor system.
  The reliability and internal consistency of the FDI (Cronbach's alpha coefficient) was 0.83 for the complete scale. Intra-class correlation was 0.79 (95% CI: 0.71-0.85) and 0.85 (95% CI: 0.78-0.89) for the physical and social well-being subscale
Kinovea Movement Analysis software | 3rd week
  An objective analysis of the human movement can help both clinical assessment and sports performance. Kinovea is a free 2D motion analysis software that can be used to measure kinematic parameters. The Kinovea software is a valid and reliable tool that can measure accurately at distances up to 5 m from the object and at an angle range of 90°-45°. Nevertheless, for optimum results an angle of 90° is suggested and trustworthy instrument because of strong intra rater reliability(0.98-0.99) and inter rater reliability (0.95-0.98).
  During recording, patients were asked to perform three movements as follows: first, raise the eyebrows (frontalis); second, smile with pursed lips (zygomatic); and third, pout the lips (orbicularis oris). The symmetry ratio was calculated while comparing each side of face

CONTACTS AND LOCATIONS:
Overall Officials: Saifa Zia, Principal Investigator — Riphah International University (Lahore)
Locations (1):
- DHQ, Kasur (Baba Bulleh Shah Hospital, District Kasur)., Kasur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardoso JR, Teixeira EC, Moreira MD, Favero FM, Fontes SV, Bulle de Oliveira AS. Effects of exercises on Bell's palsy: systematic review of randomized controlled trials. Otol Neurotol. 2008 Jun;29(4):557-60. doi: 10.1097/MAO.0b013e31816c7bf1. PMID 18520590
- [Background] Paolucci T, Cardarola A, Colonnelli P, Ferracuti G, Gonnella R, Murgia M, Santilli V, Paoloni M, Bernetti A, Agostini F, Mangone M. Give me a kiss! An integrative rehabilitative training program with motor imagery and mirror therapy for recovery of facial palsy. Eur J Phys Rehabil Med. 2020 Feb;56(1):58-67. doi: 10.23736/S1973-9087.19.05757-5. Epub 2019 Mar 27. PMID 30916916